CLINICAL TRIAL: NCT04225507
Title: Technology-Supported Treatment of Sleep Apnea in Prediabetes
Acronym: TECH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Northwestern University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB19-1445; R01DK120312 (NIH)
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-07

CONDITIONS: Sleep Apnea; PreDiabetes; Overweight or Obesity
MeSH Terms: conditions — Sleep Apnea Syndromes; Prediabetic State; Overweight; Obesity | interventions — Diet; Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Intervention (Other): Diet and exercise.
  Interventions: Behavioral: Diet and exercise coaching
- Lifestyle Plus CPAP Intervention (Experimental): CPAP treatment, diet and exercise.
  Interventions: Behavioral: Diet and exercise coaching; Other: CPAP Treatment

INTERVENTIONS:
Behavioral: Diet and exercise coaching — All participants will receive diet and exercise goals and coaching.
Other: CPAP Treatment — CPAP treatment for sleep apnea and CPAP education and adherence coaching.
  Arms: Lifestyle Plus CPAP Intervention

SUMMARY:
Despite the efficacy of intensive lifestyle interventions in prediabetes, the incidence of diabetes is rising, and thus there is a critical need for additional strategies to prevent diabetes and to reduce its cardiovascular complications in this high-risk population. Sleep apnea is a highly common condition in prediabetes, but it has been mostly ignored and undertreated in current practice. The proposed study will be the first to assess whether adding CPAP (continuous positive air pressure) treatment to a lifestyle intervention improves cardiometabolic outcomes beyond that achieved with lifestyle alone (i.e. current standard of care) in high-risk individuals with prediabetes.

DETAILED DESCRIPTION:
This is a 6-month randomized controlled, parallel group trial with two arms. After baseline, the subjects will be randomized to lifestyle intervention alone (lifestyle group) or lifestyle plus CPAP intervention (lifestyle plus CPAP group). The same metabolic and cardiovascular assessments will be performed at baseline and after 6-months of intervention.

The lifestyle group will aim to achieve a weight loss through diet and exercise. The lifestyle plus CPAP group will additionally receive CPAP treatment. All subjects will use a custom smartphone app to track weight loss and/or CPAP goals and will receive weekly coaching phone calls to maximize treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese
* Prediabetes
* Sleep apnea

Exclusion Criteria:

* Diabetic
* enrolled in a formal weight loss program
* Any underlying disease likely to limit life span and/or increase risk of interventions

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline 2-hour glucose levels at 6 months | Baseline and at 6 months
  Glucose levels will be measured at time=120min during oral glucose tolerance test

SECONDARY OUTCOMES:
Change from baseline morning blood pressure at 6 months | Baseline and 6 months
  Morning blood pressure will be measured with a blood pressure cuff while sitting

CONTACTS AND LOCATIONS:
Overall Officials: Esra Tasali, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States